CLINICAL TRIAL: NCT01767675
Title: A Phase II Randomized Study: Outcomes After Secondary Cytoreductive Surgery With or Without Carboplatin Hyperthermic Intraperitoneal Chemotherapy (HIPEC) Followed by Systemic Combination Chemotherapy for Recurrent Platinum-Sensitive Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Brief Title: Outcomes After Secondary Cytoreductive Surgery With or Without Carboplatin Hyperthermic Intraperitoneal Chemotherapy (HIPEC) Followed by Systemic Combination Chemotherapy for Recurrent Platinum-Sensitive Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Mayo Clinic (Other); Baptist Health South Florida (Other); Hartford HealthCare (Other); University of Pittsburgh (Other); University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-275
Record Dates: First submitted 2013-01-10; First posted 2013-01-14 (Estimated); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Ovarian Cancer; Fallopian Tubes Cancer; Peritoneal Cancer
Keywords: Secondary Cytoreductive Surgery; Carboplatin; Hyperthermic Intraperitoneal Chemotherapy (HIPEC); 12-275
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms

ARMS (2):
- Secondary Cytoreductive Surgery with HIPEC (Experimental): secondary cytoreductive surgery (CRS) with or without carboplatin-based hyperthermic intraperitoneal chemotherapy (HIPEC) followed by systemic combination chemotherapy for recurrent platinum-sensitive ovarian, fallopian tube, or primary peritoneal cancer. Patients will be randomized intraoperatively to undergo CRS with HIPEC (arm A) or CRS only (arm B) in a manner 1:1. Both arms will receive a standard platinum-based systemic chemotherapy postoperatively (5 cycles in arm A and 6 cycles in arm B). In some patients randomized to HIPEC at MSKCC only , peritoneal fluid and blood samples will be drawn before, during and after the HIPEC procedure.
  Interventions: Procedure: Secondary Cytoreductive Surgery; Drug: Carboplatin Hyperthermic Intraperitoneal Chemotherapy (HIPEC); Drug: platinum-based systemic chemotherapy postoperatively
- Secondary Cytoreductive Surgery without HIPEC (Experimental): secondary cytoreductive surgery (CRS) with or without carboplatin-based hyperthermic intraperitoneal chemotherapy (HIPEC) followed by systemic combination chemotherapy for recurrent platinum-sensitive ovarian, fallopian tube, or primary peritoneal cancer. Patients will be randomized intraoperatively to undergo CRS with HIPEC (arm A) or CRS only (arm B) in a manner 1:1. Both arms will receive a standard platinum-based systemic chemotherapy postoperatively (5 cycles in arm A and 6 cycles in arm B).
  Interventions: Procedure: Secondary Cytoreductive Surgery; Drug: platinum-based systemic chemotherapy postoperatively

INTERVENTIONS:
Procedure: Secondary Cytoreductive Surgery
Drug: Carboplatin Hyperthermic Intraperitoneal Chemotherapy (HIPEC)
  Arms: Secondary Cytoreductive Surgery with HIPEC
Drug: platinum-based systemic chemotherapy postoperatively — 5 cycles
  Arms: Secondary Cytoreductive Surgery with HIPEC
Drug: platinum-based systemic chemotherapy postoperatively — 6 cycles
  Arms: Secondary Cytoreductive Surgery without HIPEC

SUMMARY:
The purpose of this study is to see if the investigators can improve the treatment of this type of cancer. They want to find out what effects, good and/or bad, giving heated chemotherapy into the belly, known as hyperthermic intraperitoneal chemotherapy (HIPEC), has on the patient and this type of cancer.

The goal of HIPEC is to expose any cancer left in the abdomen after surgery to high doses of chemotherapy. The chemotherapy is heated in the hope that this will make it easier for it to get into and kill the cancer cells. The drug used for HIPEC will be carboplatin, a Food and Drug Administration (FDA) approved drug for use in ovarian, fallopian tube or primary peritoneal cancer.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Eligibility Prior to Surgery:

* Age ≥ 21 years old.
* Patients with histologic diagnosis of epithelial ovarian carcinoma, primary peritoneal carcinoma, or fallopian tube carcinoma that has recurred >6 months since platinum-based chemotherapy (first recurrence) and who are scheduled for secondary surgical evaluation/cytoreduction.
* Histologic epithelial cell types include serous, endometrioid, clear cell, or undifferentiated carcinomas, transitional cell carcinoma, mixed epithelial carcinoma, malignant Brenner's tumor, or adenocarcinoma N.O.S.
* Karnofsky Performance Status (KPS) of ≥ 70%.
* Disease-free interval ≤ 30 months.
* No prior chemotherapy in the recurrent setting. Prior hormonal therapy is permitted. Concomitant anti-neoplastic anti-hormonal therapy (including tamoxifen, aromatase inhibitors etc.) is not allowed for patients participating in study treatment. Low-dose (physiologic) estrogen hormone-replacement therapy (HRT) may be given.
* Patients receiving maintenance biologic therapy are eligible, provided their recurrence is documented more than 6 months from completion of primary cytotoxic chemotherapy (includes maintenance chemotherapy) and a minimum of 3 weeks has elapsed since their last infusion of biologic therapy at the start of protocol intervention, day 1.
* Patients must be, after evaluation by the investigator, appropriate candidates for the administration of 5 to 6 cycles of standard platinum-based combination chemotherapy (carboplatin and paclitaxel, carboplatin and liposomal doxorubicin, or carboplatin and gemcitabine) following CRS with or without HIPEC.
* Bone marrow function:
* Hemoglobin ≥ 8.5 g/dL.
* Absolute neutrophil count (ANC) ≥ 1,000/mm3.
* Platelets ≥ 100,000/mm3.
* Renal function:
* Creatinine ≤ 1.5mg/dl
* Hepatic function:
* Bilirubin ≤ 1.5 times ULN.
* ALT ≤ 3 times the ULN.
* AST ≤ 3 times the ULN.
* Neurologic function:
* Peripheral neuropathy ≤ CTC AE grade 2.
* Blood coagulation parameters:
* PT with an INR of ≤ 1.5 and a PTT ≤ 1.5 times the ULN. For patients on full-dose oral anti-coagulation (such as warfarin or rivaroxaban), in-range INR (usually between 2 and 3) and a PTT <1.2 times the ULN.
* Patients of childbearing potential must have a negative serum pregnancy test within 2 weeks prior to CRS and must be practicing an effective form of contraception during the study period.

Inclusion Criteria for Eligibility Post-Surgery:

* Patients will be consented prior to the surgical evaluation/cytoreductive surgery. Patients must have less than or equal to 0.5cm residual disease at the completion of the secondary surgery to be eligible for the study.

Exclusion Criteria:

Exclusion Criteria for Eligibility Prior to Surgery:

* Tumors of low malignant potential (borderline carcinomas).
* Subjects who have received prior radiotherapy to any portion of the abdominal cavity or pelvis are excluded.
* Patients with a history of primary endometrial cancer are excluded unless the following conditions are met:
* Stage not greater than IA.
* Not a poorly differentiated subtype (including papillary serous, clear cell or other FIGO grade 3 lesions)
* With the exception of non-melanoma skin cancer and other specific malignancies as noted above, subjects with other invasive malignancies, who had any evidence of the other cancer present within the last 1 year or whose previous cancer treatment contraindicates this protocol therapy, are excluded.
* Subjects with known active acute hepatitis.
* Subjects with active infection that requires parenteral antibiotics.
* Active coronary artery disease (defined as unstable angina or a positive cardiac stress test).
* Patients with a history of coronary artery disease may be included if they have had a normal stress test within 30 days of enrollment.
* Uncontrolled hypertension defined as > 140/90 and not cleared for surgery at the time of consent..
* New York Heart Association (NYHA) Class II or higher Congestive heart failure.
* History of cerebrovascular disease.
* Immune deficiency: Clinically significant primary or acquired immune deficiency (i.e. AIDS or on immunosuppressive medication after organ transplant).
* Patients with other concurrent severe medical problems unrelated to the malignancy that would significantly limit full compliance with the study or places them at an unacceptable risk for participation in the study.
* Patients with known carboplatin or cisplatin allergy.
* Life expectancy < 12 weeks.

Exclusion Criteria for Eligibility Post-Surgery:

* Evidence of extensive intraperitoneal adhesions at the time of surgery, as determined by the operating surgeon which prohibits intraperitoneal therapy.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2013-01-08 (Actual); Primary Completion 2025-08-26 (Actual); Study Completion 2025-08-26 (Actual)

PRIMARY OUTCOMES:
determine the proportion of patients who are without evidence of disease progression | 24 months
  A proportion of patients ≥ 40%, who are without evidence of disease progression at 24 months, is considered acceptable, whereas a proportion of ≤ 25% is considered not acceptable in this patient population.

SECONDARY OUTCOMES:
To determine the toxicity and postoperative complications rate | 4 weeks post op
  The safety endpoint of our trial is to determine toxicity and postoperative complication rates in both arms using NCI Common Terminology Criteria for Adverse Events version 4.0. and MSKCC Surgical Secondary Events Grading System for complications.
determine the completion rate of four cycles | 5 years
  A secondary analysis of estimating the completion rate will be conducted. The completion rate and a 95% confidence interval will be calculated for each arm separately. Completion is defined as patients being able to complete ≥ 4 out of 5 or 6 cycles of a standard systemic chemotherapy.
pharmacokinetics | 5 years
  in a subset of patients randomized to receive HIPEC in the OR. In patients randomized to HIPEC, peritoneal fluid and blood samples only from MSKCC patients will be drawn before, during and after the HIPEC procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Chi, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (11):
- United States (11):
  - Hartford Healthcare Cancer Institute @ Hartford Hospital, Hartford, Connecticut
  - Baptist Health South Florida, Miami, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (All protocol activities, except surgery), Uniondale, New York

REFERENCES:
- [Derived] Zivanovic O, Chi DS, Zhou Q, Iasonos A, Konner JA, Makker V, Grisham RN, Brown AK, Nerenstone S, Diaz JP, Schroeder ED, Langstraat CL, Paroder V, Lakhman Y, Soldan K, Su K, Gardner GJ, Andikyan V, Guo J, Jewell EL, Long Roche K, Troso-Sandoval T, Lichtman SM, Moukarzel LA, Dessources K, Abu-Rustum NR, Aghajanian C, Tew WP, Beumer J, Sonoda Y, O'Cearbhaill RE. Secondary Cytoreduction and Carboplatin Hyperthermic Intraperitoneal Chemotherapy for Platinum-Sensitive Recurrent Ovarian Cancer: An MSK Team Ovary Phase II Study. J Clin Oncol. 2021 Aug 10;39(23):2594-2604. doi: 10.1200/JCO.21.00605. Epub 2021 May 21. PMID 34019431
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/